CLINICAL TRIAL: NCT05208008
Title: on the Daily Activity, Sleep Pattern, and Stress Level of Military Veterans With PTSD
Brief Title: Effect of Owning a Service Dog on Military Veterans With PTSD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ANIMAL CONTACT 3
Record Dates: First submitted 2021-12-20; First posted 2022-01-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Physiological Responses; Sleep Disorders, Circadian Rhythm; Stress, Emotional
Keywords: Human-animal contact; Non-invasive measure
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With service dog: Veterans living with a certified service dog
  Interventions: Other: With service dog
- Without service dog: Veterans living without a certified service dog

INTERVENTIONS:
Other: With service dog — No intervention
  Groups: With service dog

SUMMARY:
The study aims to investigate the effects of a service dog on military veterans with post traumatic stress syndrome (PTSD). The investigators will use non-invasive measures of the physiological responses, data obtained via dairy keeping, accelerometer data estimating activity and sleep patterns, and baseline information including psychological measures validated for this specific population.

DETAILED DESCRIPTION:
The investigators will measure and compare the immediate effect of the presence of the dog, on days with low stress and high stress, using non-invasive measures of the physiological response, diary notes, and data on activity and sleep pattern The latter will also be collected for the service dogs. The investigators will apply a cross-sectional design. The participants will be divided into two groups based on whether they own a certified service dog (treatment group) or are on a waitlist for a service dog (control group).

The experimental period will consist of a 14-day period. In the preceding week the participants receive a visit, where they will be given instructions to fill in a diary, how to collect and store saliva samples, and use equipment for data collection. In the diary they record their daily activities and any situation perceived to be stressful during the experimental period. In the experimental period, the participants will wear an accelerometer. Every second day, the particpants will wear equipment measuring their heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Have been deployed in a war zone
* Fulfil criteria for PTSD
* Fulfil criteria for receiving a certified service dog
* If having a service dog, they must have owned the dog for more than 6 months, and the dog must be at leat 2 years of age

Exclusion Criteria:

* Use of alcohol or drugs to an extent that it affects the ability to attend to ordinary daily activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Military veterans, that either already ave a certified service dog, or are approved to receive a certified service dog, but on a waitlist.
  Furthermore, the military veterans should fulfill the inclusion criteria.
  The are recruited with help from the Danish Military, and the initial contact is established when potential participants respond to the advertisements by contacting of the scientific staff of the project.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily activity pattern | In the experimental period, which is 14 days
  Daily activity pattern measured with a wrist-worn accelerometer
Sleep pattern | In the experimental period, which is 14 days
  Sleep pattern measured with a wrist-worn accelerometer
Salivary, Cortisol | Day 1 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 1 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 2 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 2 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 3 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 3 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 4 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 4 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 5 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 5 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 6 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 6 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 7 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 7 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 8 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 8 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 9 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 9 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 10 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 10 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 11 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 11 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 12 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 12 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 13 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 13 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 14 of the experimental period at 11 a.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary, Cortisol | Day 14 of the experimental period at 8 p.m.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Blood pressure | Day 1 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 1 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 2 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 2 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 3 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 3 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 4 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 4 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 5 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 5 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 6 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 6 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 7 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 7 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 8 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 8 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 9 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 9 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 10 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 10 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 11 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 11 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 12 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 12 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 13 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 13 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 14 of the experimental period at 11 a.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Blood pressure | Day 14 of the experimental period at 8 p.m.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Heart rate | Day 2 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate | Day 4 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate | Day 6 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate | Day 8 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate | Day 10 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate | Day 12 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate | Day 14 of the experimental period
  The test person wears either self-adhesive electrodes or a belt around their chest and the heart rate is measured non-invasively
Heart rate variability | Day 2 of the experimental period
  Heart rate variability is calculated from heart rate data
Heart rate variability | Day 4 of the experimental period
  Heart rate variability is calculated from heart rate data
Heart rate variability | Day 6 of the experimental period
  Heart rate variability is calculated from heart rate data
Heart rate variability | Day 8 of the experimental period
  Heart rate variability is calculated from heart rate data
Heart rate variability | Day 10 of the experimental period
  Heart rate variability is calculated from heart rate data
Heart rate variability | Day 12 of the experimental period
  Heart rate variability is calculated from heart rate data
Heart rate variability | Day 14 of the experimental period
  Heart rate variability is calculated from heart rate data
Dairy notes regarding stressful events | Day 1 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 2 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 3 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 4 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 5 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 6 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 7 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 8 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 9 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 10 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 11 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 12 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 13 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period
Dairy notes regarding stressful events | Day 14 of the experimental period
  The participant notes whether any situations, perceived to be stressful has happened, during each of the 14 days in the experimental peiod.during the experimental period

CONTACTS AND LOCATIONS:
Locations (1):
- Karen Thodberg, Højslev, Denmark

IPD SHARING:
Plan to Share IPD: No